CLINICAL TRIAL: NCT06933121
Title: Empowering Healthy Lifestyle Behaviour Through Personalised Intervention Portfolios to Prevent and Control Obesity in Children - UEV Pilot Study
Acronym: UEVCh_HW8
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Évora (Other)
Responsible Party: Principal Investigator, Elsa Lamy, Principal Investigator, Head of the Laboratory of Oral Biology and Salivary Proteomics, University of Évora
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UEVHeightW8Children
Record Dates: First submitted 2024-11-15; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-03

CONDITIONS: Obesity and Obesity-related Medical Conditions
Keywords: Obesity; Overweight; Prevention; Digital-twin; Lifestyle
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Intervention Model Description: In this short-term study, the intervention with a digital solution, with personalized recommendations about lifestyle aspects, will be used to all participants. Data collection will be made at the beginning and at the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Digital intervention group (Experimental): Group of individuals that will have access to the digital tool and that will be followed for their used and efficacy.
  Interventions: Device: Digital twin for personalized recommendations

INTERVENTIONS:
Device: Digital twin for personalized recommendations — The intervention is the developed eHealth solution, i.e. the healthy lifestyle recommender system. It is based on a previously developed meal recommender system, but will be much extended, resulting in a multilevel portfolio intervention regarding:
  1. Suggesting personalized meal recommendations,
  2. Proposing physical activities tailored to the individuals' capabilities and preferences,
  3. Measuring and considering emotional and psychological parameters,
  4. Proposing additional healthy life-style patterns regarding e.g. sleeping patterns, alcohol and tobacco consumption, engaging in social activities etc.
  The detailed nature of the interventions will first be developed during co-creation and then targeted to the participating individual. Moreover, particular attention will be given, since this needs to be a eHealth solution easy to be used by children. The intervention will include collecting urine and saliva samples, as well as measuring anthropometrics and collecting data (persona

SUMMARY:
This study is being performed under the European Consortium HealthyW8 that has the main objective of developing a digital tool for personalized recommendations for healthy lifestyle and prevention of obesity. This human study will be a pilot trial that will precede a planned more long-term intervention trial. It will focus on children (age 5 to 12 y) and parents. The main purpose is to study whether the healthy lifestyle recommender solution, reflecting a multi-portfolio intervention and developed within this project, is well accepted by the participants, has a decent adherence (i.e. user time of the app), and whether the overall design is well suited to the participants, in order that they will improve dietary habits. This study will be of longitudinal design without a control group.

DETAILED DESCRIPTION:
At present, numbers of persons with overweight and obesity continue to grow in most countries worldwide. Children and young adults are at risk for different reasons: in the case of children, dietary habits and lifestyle is starting to be developed and if, at this phase, children do not acquire healthy habits, it will be probable that they will have a higher potential to develop obesity and the associated co-morbidities. It is at this stage that food preferences develop. Moreover, children obesity is increasing and it is known that an obese or pre-obese children will have a higher propensity to be an obese adult. For young adults, the risks and concerns are different. Is in this period of life that most people starts an independent life, and consequently decide their food and lifestyle choices, with an increase in irregularity of meals and unhealthy food choices, together with changes in physical activity habits and social or individual pressures. It is essential to give them tools that will allow them to make healthy choices and to have healthy habits, since they will be the future adult population that will raise and inspire the next generation. As solutions to combat the trend toward increasing overweight and obesity are much in need, the present study aims to intervene with the developed healthy lifestyle recommender solution to address various factors known to constitute a risk for developing obesity, including socio-demographic aspects, psychological/behavioural ones, physical activity, dietary patterns, among other. Such a multi-dimensional portfolio approach is believed to be very much needed for the prevention of obesity and co-morbidities, and the personalization of the solution, as well as the nudging/gamification aspects will strive to ensure a high long-term adherence to the developed solution.

The primary objective of the study is to determine whether the developed healthy-lifestyle recommender solution can be successfully applied to the target population (children and their parents), and whether they adhere to using it frequently during the duration of the study.

This will be assessed by adherence time to the lifestyle recommender solution and questionnaires addressing the user-friendliness and limitation or problems encountered. Secondly, the investigators will study whether the assessment of endpoints required for the ensuing long-term study can be well assessed within the study and if despite the limited time of the intervention duration, the intervention will be able to improve some markers related to the risk of obesity and associated co-morbidities.

ELIGIBILITY:
Inclusion Criteria:

* Children (age 5-12 y) and, at least, one of their parents
* To reside in Portugal (for logistic reasons)
* To be overweight (BMI percentile > 85%)
* Both boys and girls

Exclusion Criteria:

* To have manifest chronic diseases (e.g. cancer)
* To be already in energy restriction or following a specific diet (on their own or advised by their physician)
* To have eating behaviour pathologies

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-04-14 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Adherence to digital tool | At the end of the study, after 3-month intervention.
  Adherence time to the lifestyle recommender solution and questionnaires addressing the user-friendliness and limitation or problems encountered. This will be quantified according to the scale of the questionnaires.

SECONDARY OUTCOMES:
Changes in BMI | 3-months
  we will study whether the assessment of endpoints required for the ensuing long-term study can be well assessed within the study and if despite the limited time of the intervention duration, the intervention will be able to improve some markers related to the risk of obesity and associated co-morbidities. Toward this end, change of BMI, relatively to the beginning of the intervention will be assessed.
Salivary biomarkers of stress | 3-months
  The investigators will study how the intervention will be able to change salivary cortisol and alpha-amylase concentrations.
Salivary biomarkers of physiology and metabolism | 3-months
  The levels of different salivary molecules will be measured in the periods before and after intervention, namely: salivary glucose and insulin, salivary C-reactive protein - CRP concentrations.
Dietary habits | At the beginning of the study
  The dietary habits of children, at the beginning of the study, will be determined through validated Food Frequency Questionnaires, which will allow to quantify the average amount of each food type consumed per day, as well as the amounts of macro- and micronutrients consumed per day.

IPD SHARING:
Plan to Share IPD: No
Individual data will be not shared. Data will be treated and only treated data will be available. Only the PI of the study will be access to the correspondence between participant identification and codification that will be given to each participant. There is no need of having identification of participants to reach the conclusions about the study.

REFERENCES:
- See also: Website of HealthyW8 project, with detailed description about aims, consortium and project. — https://www.healthyw8.eu